CLINICAL TRIAL: NCT00266149
Title: Phase 3: Metabolism of Lamotrigine During Treatment With Oral Contraceptives
Brief Title: Lamotrigine and Oral Contraceptives
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LMS: j.nr. 2612-2188; EK:j. nr. 20030009
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2005-12

CONDITIONS: Epilepsy
Keywords: Pharmacokinetics; Lamotrigine; Oral Contraceptives; UGT; Glucuronidation.
MeSH Terms: conditions — Epilepsy | interventions — Contraceptives, Oral; Lamotrigine

INTERVENTIONS:
Drug: Oral contraception
Drug: Lamotrigine

SUMMARY:
The present study evaluates the effect of oral contraceptives on lamotrigine plasma concentrations in a double blind, placebo controlled, cross-over study in patients with epilepsy.

DETAILED DESCRIPTION:
Lamotrigine is widely used as an antiepileptic drug in the treatment of newly onset as well as refractory epilepsy (1;2). Lamotrigine is unique among the antiepileptic drug since the major route (76%) of elimination is conjugation with glucuronic acid (glucuronidation) (3). This conjugation reaction is catalyzed by the uridine 5'-diphosphate (UDP)-glucuronosyltransferases (UGTs); of which the isoform UGT1A4 probably is the major route of metabolism in humans (3). The pathway is inhibited by valproate and induced by other anticonvulsants (3), and explains the effect of these drugs on lamotrgine metabolism (4). Other drugs that are metabolized via direct glucoronidation may interfere with the metabolism of lamotrigine e.g. acetaminophen (5). Estrogeneous substrates are metabolized via glucuronidation (6-8) and may potentially interact with the metabolism of lamotrigine. In the development of lamotrigine for use in epilepsy patients the effect on the oral contraceptive pill was studied. In contrast to other commonly used antiepileptic drugs e.g. carbamazepine and phenytoin(9), lamotrigine did not significantly influence the constituents of the oral contraceptive pill (10-12). In addition, it was initially assumed from population pharmacokinetic studies, that oral contraceptives did not influence the metabolism of lamotrigine (13).However, recent retrospective studies indicate that oral contraceptives may increase the metabolism of lamotrigine resulting in a significant decrease in plasma concentration of lamotrigine when given with oral contraceptives (14;15). This effect is probably related to the ethinyl estradiol content of the combined contracetive pill and no the progesterone content (16).

To confirm and further extend these findings, the present study evaluates the effect of oral contraceptives on lamotrigine plasma concentrations in a double blind, placebo controlled, cross-over study in patients with epilepsy.

Reference List

1. French JA, Kanner AM, Bautista J, Abou-Khalil B, Browne T, Harden CL et al. Efficacy and Tolerability of the New Antiepileptic Drugs, II: Treatment of Refractory Epilepsy: Report of the TTA and QSS Subcommittees of the American Academy of Neurology and the American Epilepsy Society. Epilepsia 2004; 45(5):410-423.
2. French JA, Kanner AM, Bautista J, Abou-Khalil B, Browne T, Harden CL et al. Efficacy and Tolerability of the New Antiepileptic Drugs, I: Treatment of New-Onset Epilepsy: Report of the TTA and QSS Subcommittees of the American Academy of Neurology and the American Epilepsy Society. Epilepsia 2004; 45(5):401-409.
3. Dickins M, Chen C. Lamotrigine. Chemistry, Biotransformation and Pharmacokinetics. In: Levy RH, Mattson RH, Meldrum BS, Perucca E, editors. Antiepileptic Drugs. Philidelphia: Lippincott, Williams & Wilkins, 2002: 370-379.
4. Patsalos PN, Perucca E. Clinically important drug interactions in epilepsy: general features and interactions between antiepileptic drugs. Lancet Neurol 2003; 2(6):347-356.
5. Depot M, Powell JR, Messenheimer JAJ, Cloutier G, Dalton MJ. Kinetic effects of multiple oral doses of acetaminophen on a single oral dose of lamotrigine. Clin Pharmacol Ther 1990; 48(4):346-355.
6. Tephly TR, Green MD. UDP-Glucuronosyltransferases. In: Levy RH, Thummel KE, Trager W, Hansten PD, Eichelbaum M, editors. Metabolic Drug Interactions. Philidelphia: Lippincott, Williams & Wilkins, 2000: 161-174.
7. Shipkova M, Wieland E. Glucuronidation in therapeutic drug monitoring. Clin Chim Acta 2005; 358(1-2):2-23.
8. Ebner T, Remmel RP, Burchell B. Human bilirubin UDP-glucuronosyltransferase catalyzes the glucuronidation of ethinylestradiol. Mol Pharmacol 1993; 43(4):649-654.
9. Patsalos PN, Perucca E. Clinically important drug interactions in epilepsy: interactions between antiepileptic drugs and other drugs. Lancet Neurol 2003; 2(8):473-481.
10. Crawford P. Interactions between antiepileptic drugs and hormonal contraception. CNS Drugs 2002 ;16 (4 ):263 -72 2002; 16(4):263-272.
11. Doose DR, Wang SS, Padmanabhan M, Schwabe S, Jacobs D, Bialer M. Effect of topiramate or carbamazepine on the pharmacokinetics of an oral contraceptive containing norethindrone and ethinyl estradiol in healthy obese and nonobese female subjects. Epilepsia 2003 Apr ;44 (4 ):540 -9 44(4):540-549.
12. Holdish T, Whiteman P, Orme M, Back D, Ward S. Effect of lamotrigine on the pharmacology of the combined oral contraceptive pill. Epilepsia 32[suppl. 1], s96. 1991.
13. Hussein Z, Posner J. Population pharmacokinetics of lamotrigine monotherapy in patients with epilepsy: retrospective analysis of routine monitoring data. Br J Clin Pharmacol 1997; 43(5):457-465.
14. Sabers A, Ohman I, Christensen J, Tomson T. Oral contraceptives reduce lamotrigine plasma levels. Neurology 2003 Aug 26 ;61 (4 ):570 -1 2003; 61(4):570-571.
15. Sabers A, Buchholt JM, ULDALL P, Hansen EL. Lamotrigine plasma levels reduced by oral contraceptives. Epilepsy Res 2001 Nov ;47 (1 -2 ):151 -4 47(1-2):151-154.
16. Reimers A, Helde G, Brodtkorb E. Ethinyl estradiol, not progestogens, reduces lamotrigine serum concentrations. Epilepsia 2005; 46(9):1414-1417.

ELIGIBILITY:
Inclusion Criteria:

Women with epilepsy, treated with lamotrigine in monotherapy and taking combination type oral contraceptives, and who were between 18 and 40 years of age, were candidates for inclusion in the study. Patients should agree to use contraception of barrier type throughout the study (see study design).

Exclusion Criteria:

Patients were not admitted to the study if any of the following criteria were present: (1) pregnancy, (2) breastfeeding, (3) affected liver function, (4) affected kidney function, (5) daily intake of drugs with known or suspected influence on the metabolism of lamotrigine (acetaminophen and sertralin).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10
Dates: Start 2003-06; Study Completion 2005-05

PRIMARY OUTCOMES:
The dose corrected trough concentration of lamotrigine following 21 days of placebo treatment compared to the dose

SECONDARY OUTCOMES:
Secondary endpoints; the trough concentration of lamotrigine following 7 days of pause with the oral contraceptive pill, and the proportion of lamotrigine to lamotrigine metabolites found in urine samples following treatment with placebo and the o

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Christensen, MD, PhD, Principal Investigator — Department of Neurology, Aarhus University Hospital, 8000 Aarhus C
Locations (1):
- Department of Neurology, Aarhus University Hospital, Aarhus, Aarhus, Denmark

REFERENCES:
- [Background] French JA, Kanner AM, Bautista J, Abou-Khalil B, Browne T, Harden CL, Theodore WH, Bazil C, Stern J, Schachter SC, Bergen D, Hirtz D, Montouris GD, Nespeca M, Gidal B, Marks WJ Jr, Turk WR, Fischer JH, Bourgeois B, Wilner A, Faught RE Jr, Sachdeo RC, Beydoun A, Glauser TA; American Academy of Neurology Therapeutics and Technology Assessment Subcommittee; American Academy of Neurology Quality Standards Subcommittee; American Epilepsy Society Therapeutics and Technology Assessment Subcommittee; American Epilepsy Society Quality Standards Subcommittee. Efficacy and tolerability of the new antiepileptic drugs, II: Treatment of refractory epilepsy: report of the TTA and QSS Subcommittees of the American Academy of Neurology and the American Epilepsy Society. Epilepsia. 2004 May;45(5):410-23. doi: 10.1111/j.0013-9580.2004.06304.x. PMID 15101822
- [Background] French JA, Kanner AM, Bautista J, Abou-Khalil B, Browne T, Harden CL, Theodore WH, Bazil C, Stern J, Schachter SC, Bergen D, Hirtz D, Montouris GD, Nespeca M, Gidal B, Marks WJ Jr, Turk WR, Fischer JH, Bourgeois B, Wilner A, Faught RE Jr, Sachdeo RC, Beydoun A, Glauser TA; American Academy of Neurology Therapeutics and Technology Assessment Subcommittee; American Academy of Neurology Quality Standards Subcommittee; American Epilepsy Society Quality Standards Subcommittee; American Epilepsy Society Therapeutics and Technology Assessment Subcommittee. Efficacy and tolerability of the new antiepileptic drugs, I: Treatment of new-onset epilepsy: report of the TTA and QSS Subcommittees of the American Academy of Neurology and the American Epilepsy Society. Epilepsia. 2004 May;45(5):401-9. doi: 10.1111/j.0013-9580.2004.06204.x. PMID 15101821
- [Background] Patsalos PN, Perucca E. Clinically important drug interactions in epilepsy: general features and interactions between antiepileptic drugs. Lancet Neurol. 2003 Jun;2(6):347-56. doi: 10.1016/s1474-4422(03)00409-5. PMID 12849151
- [Background] Depot M, Powell JR, Messenheimer JA Jr, Cloutier G, Dalton MJ. Kinetic effects of multiple oral doses of acetaminophen on a single oral dose of lamotrigine. Clin Pharmacol Ther. 1990 Oct;48(4):346-55. doi: 10.1038/clpt.1990.162. PMID 2225696
- [Background] Shipkova M, Wieland E. Glucuronidation in therapeutic drug monitoring. Clin Chim Acta. 2005 Aug;358(1-2):2-23. doi: 10.1016/j.cccn.2005.02.023. PMID 15893300
- See also: Danish Medicines Agency — http://www.dkma.dk